CLINICAL TRIAL: NCT04683081
Title: Cervical Ripening: a Comparison of Three Mechanical Methods in Term of Patient Satisfaction
Brief Title: Patient Satisfaction With Mechanical Cervical Ripening
Status: Completed | Type: Observational
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kemal Sarsmaz, MD, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Other Study IDs: patient satisfaction
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Satisfaction, Patient
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Foley catheter group: pregnant women who were applied Foley catheter for cervical ripening
  Interventions: Device: mechanical cervical ripening
- Cook balloon catheter group: pregnant women who were applied Cook balloon catheter for cervical ripening
  Interventions: Device: mechanical cervical ripening
- Modified double-balloon Foley catheter group: pregnant women who were applied modified double-balloon Foley catheter for cervical ripening
  Interventions: Device: mechanical cervical ripening

INTERVENTIONS:
Device: mechanical cervical ripening — mechanical cervical ripening methods have been used to make the cervix more eligible for vaginal delivery

SUMMARY:
In this study, we aimed to compare three mechanical methods such as foley catheter, cook balloon catheter and modified double-balloon Foley catheter for cervical ripening in terms of patient satisfaction

DETAILED DESCRIPTION:
This is a prospective observational study. The planned sample size is 34 pregnant women per group with 90% power and 0.05 alpha error.

VAS score systems and Salmon's item list were used to evaluate the satisfaction level.

The inclusion criteria are age between 18 and 40, singleton pregnancy, vertex presentation, bishop score <6, using a foley catheter cook balloon catheter or modified double-balloon Foley catheter for cervical ripening and high-risk pregnancy (Oligohydramnios, polyhydramnios, intrauterine growth retardation, pregestational or gestational diabetes, hypertensive disorders).

The exclusion criteria are being younger than 18 or over 40, communication problems, bishop score >6, being at active labor, multifetal pregnancy, non-vertex presentation, scarred uterus (cesarean or myomectomy), known fetal structural or chromosomal anomaly, presence of non-reassuring fetal cardiotocography before cervical ripening, regional anesthesia during the first stage, operative delivery, presence of maternal, fetal or neonatal complication.

The primary outcomes are the differences in satisfaction level between methods with using either the VAS score system or Salmon's item list and pain scores.

The secondary outcomes are the effects of giving birth within 24 hours, parity status, the length of the first stage of labor education level and cesarean section due to failed induction on the satisfaction level.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40
* Singleton pregnancy
* Vertex presentation
* Bishop score <6
* Using a Foley catheter cook balloon catheter or modified double-balloon Foley catheter for cervical ripening
* High-risk pregnancy (Oligohydramnios, polyhydramnios, intrauterine growth retardation, pregestational or gestational diabetes, hypertensive disorders).

Exclusion Criteria:

* Being younger than 18 or over 40
* Communication problems
* Bishop score >6
* Being at active labor
* Multifetal pregnancy
* Non-vertex presentation
* Scarred uterus (cesarean or myomectomy)
* Known fetal structural or chromosomal anomaly
* Presence of non-reassuring fetal cardiotocography before cervical ripening
* Regional anesthesia during the first stage
* Operative delivery
* Presence of maternal, fetal or neonatal complication.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who were applied one of the mechanical cervical ripening methods, Foley catheter, Cook balloon catheter or modified double-balloon Foley catheter
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction level | within the first 24 hours after birth
  Overall patient satisfaction score is obteined by VAS score system and Salmon's items list
Pain scores | immediately after application
  Pain scores are obteined by VAS score system

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Etlik Zubeyde Hanim Women's Health Care, Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Lim SE, Tan TL, Ng GYH, Tagore S, Kyaw EEP, Yeo GSH. Patient satisfaction with the cervical ripening balloon as a method for induction of labour: a randomised controlled trial. Singapore Med J. 2018 Aug;59(8):419-424. doi: 10.11622/smedj.2018097. PMID 30175373
- [Background] Tomlinson AJ, Archer PA, Hobson S. Induction of labour: a comparison of two methods with particular concern to patient acceptability. J Obstet Gynaecol. 2001 May;21(3):239-41. doi: 10.1080/01443610120046314. PMID 12521850
- [Background] Akca A, Corbacioglu Esmer A, Ozyurek ES, Aydin A, Korkmaz N, Gorgen H, Akbayir O. The influence of the systematic birth preparation program on childbirth satisfaction. Arch Gynecol Obstet. 2017 May;295(5):1127-1133. doi: 10.1007/s00404-017-4345-5. Epub 2017 Mar 16. PMID 28303340